CLINICAL TRIAL: NCT06086743
Title: Effects of EMS Training on Muscle Strength in Young Healthy Adults
Brief Title: Effects of EMS Training on Muscle Strength
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/MS-PT/01614 MUHAMMAD FAHAD
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Muscle Strength
Keywords: Muscle strength; Electrical Muscle stimulation; Young adults; Muscle Bulk; Strength Training
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): 10 min of warm up exercises will be performed.
  * Arm swings
  * Jogging on the spot
  * Walks on treadmill The following exercises will be performed along with EMS after warm up exercises.
  * Bicep curls
  * Triceps dips
  * Squats
  * Quadriceps chair
  The following cool down exercises will be performed after resistance exercises along with EMS.
  * Light jogging and walking
  * Upper body stretches
  * Knee to chest pose Galvanic current would be administer, with intensity of 100 A.
  Interventions: Other: Experimental Group
- Control Group (Active Comparator): 10 min of warm up exercises will be performed.
  * Arm swings
  * Jogging on the spot
  * Walks on treadmill The following exercises will be performed after warmups.
  * Bicep curls
  * Triceps dips
  * Squats
  * Quadriceps chair
  The following cool down exercises will be performed after resistance exercises.
  * Light jogging and walking
  * Upper body stretches
  * Knee to chest pose
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Experimental Group — This group will perform 10 minutes of same warm up exercises. After warm up participants will perform 4 resistance exercises with induced EMS. The assessment of muscle strength, muscle bulk and muscle fat of the participants will be carried out at baseline before resistance exercises. the intensity of EMS would be 100A and it would remain same throughout training session. The current administered would be galvanic current. Initially the weight will be adjusted according to 1 repetition maximum, and it will increase 2kg after 3 week. 3 sets of every exercise would be performed; every set will have 12 repetitions. These exercises will be performed 3 days a week for 6 weeks. Readings of both the groups will be taken at baseline and at the end of last week.
  Arms: Experimental Group
Other: Control Group — Group B (Control group)will perform 10 minutes of same warm up exercises (Arm swings, jogging on the spot, Walks on treadmill). Group B will perform same 4 resistance exercises without EMS. These 4 exercises include Bicep curls, Triceps dips, Quadriceps chair and squats.The assessment of muscle strength, muscle bulk and muscle fat of the participants will be carried out at baseline before resistance exercises and the participants will be instructed, not to perform any kind of exercise during this period.Initially the weight will be adjusted according to 1 repetition maximum, and it will increase 2kg after 3 week. 3 sets of every exercise would be performed; every set will have 12 repetitions. These exercises will be performed 3 days a week for 6 weeks. Readings of both the groups will be taken at baseline and at the end of last week.
  Arms: Control Group

SUMMARY:
The goal of this study is to determine the effects of EMS induced muscle strengthening on muscle strength and muscle bulk in young healthy adults. The main question it aims to answer is:

Will Electrical muscle stimulation significantly improve muscle strength in young adults.

The participants falling in our inclusion criteria will be given a brief description about the exercise protocol. After informed consent, the participants will be randomized into two groups: Group A (Experimental group) and group B (Control group). Both groups will perform 10 minutes of same warm up exercises (Arm swings, jogging on the spot, Walks on treadmill). After warm up exercises, the participants in Group A (Experimental group) will perform resistance exercises with induced EMS while Group B (Control group) will perform same resistance exercises without EMS.

DETAILED DESCRIPTION:
The Electrical muscle stimulation (EMS) is a popular technique in the fields of physical therapy, rehabilitation, and sports training for decades. EMS involves the use of electrical impulses to stimulate muscle contractions, which can help prevent muscle atrophy, improve blood flow to the area, and promote healing. It has also been used to increase muscle strength and endurance, making it an effective tool for rehabilitation and sports training.

Some research has suggested that EMS may improve muscle mass, but this is likely to be a result of increased muscle activation and recruitment, rather than actual muscle hypertrophy (i.e., an increase in the size of individual muscle fibers). In other words, EMS may help to strengthen existing muscle fibers and improve muscle tone, but it is unlikely to result in significant increases in muscle size

The aim of this study is to investigate the potential effects of electrical muscle stimulation (EMS) training on muscle strength in young and healthy adults. EMS involves the use of electrical impulses to stimulate muscle contractions, and it has been suggested as a time-efficient and effective method for increasing muscle strength and overall fitness. However, there is limited scientific evidence on the effectiveness of EMS training on muscle strength in young and healthy adults. Therefore, this study aims to address this gap in the literature by examining the effects of EMS training on muscle strength in this population.

ELIGIBILITY:
Inclusion Criteria:

* Male.
* 18-35 years.
* Training for more than 6 months

Exclusion Criteria:

* Any systemic disease.
* Any musculoskeletal disorder.
* Any structural deformity.
* Recent injury or trauma.
* Individuals with implanted medical devices.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 64 (Estimated)
Dates: Start 2023-08-03 (Actual); Primary Completion 2024-02-15 (Estimated); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
Muscle Strength | 6 weeks
  Dynamometer will be used in this study to measure muscle strength. A dynamometer is a device that is commonly used to measure muscle strength. It measures the maximum force that a muscle or muscle group can generate. It to measure muscle strength dynamometer has a of reliability of 0.89
Muscle Bulk | 6 weeks
  The muscle bulk will be measured by measuring tape. Measuring muscle circumference can provide an estimate of muscle size or muscle hypertrophy, which can be used to evaluate the effectiveness of interventions such as exercise or dietary changes
One Repetition maximum | 6 Weeks
  One repetition maximum (1RM) is the maximum amount of weight that a person can lift for a single repetition with good form for a specific exercise. It is often used as a measure of strength and is commonly used to prescribe resistance training programs. It has a reliability and validity of 0.64

SECONDARY OUTCOMES:
Muscle Flexibility | 6 Weeks
  Bicep flexibility can be measured using a special test called the Bicep Flexibility Test. This test is designed to assess the flexibility of the bicep muscle and the range of motion of the shoulder joint.
  Triceps flexibility can be measured through a special test called the Triceps Brachii Stretch Test. This test is commonly used in sports and fitness settings to assess the flexibility of the triceps muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Jawad Naweed, MS-SPT, Principal Investigator — Riphah International University
Locations (1):
- Chal Foundation, Balakot, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No